CLINICAL TRIAL: NCT04138420
Title: Study of Retinal and Vascular Features by Optical Coherence Tomography and Optical Coherence Tomography Angiography After Intravitreal Injections of Bevacizumab in Exudative Age-related Macular Degeneration
Brief Title: Evaluation of Retinal and Vascular Features in Macular Degeneration After Intravitreal Injections of Bevacizumab
Status: Completed | Type: Observational
Sponsor: Federico II University (Other)
Responsible Party: Principal Investigator, Gilda Cennamo, Gilda Cennamo, Federico II University
Other Study IDs: PT1124/14
Record Dates: First submitted 2019-10-19; First posted 2019-10-24 (Actual); Last update posted 2019-10-24 (Actual); Status verified 2019-10

CONDITIONS: Exudative Age-related Macular Degeneration
Keywords: optical coherence tomography angiography; optical coherence tomography angiography angiography; bevacizumab; vascular endothelial growth factor antagonists; intravitreal injection
MeSH Terms: interventions — Bevacizumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients receiving Bevacizumab: Bevacizumab, intravitreal injection, three monthly, dosage: 1.25 mg/0.05 mL.
  Interventions: Drug: Bevacizumab Injection

INTERVENTIONS:
Drug: Bevacizumab Injection — Three monthly intravitreal injections of bevacizumab (1.25 mg/0.05 mL)
  Other Names: Avastin

SUMMARY:
This study evaluates the retinal and vascular features in patients with macular degeneration under the effects of Bevacizumab intravitreal injections using optical coherence tomography and optical coherence tomography angiography.

DETAILED DESCRIPTION:
Bevacizumab is a vascular endothelial growth factor antagonist represent an efficacy treatment for exudative age-related macular degeneration acting on vascular hyperpermeability.

The optical coherence tomography and optical coherence tomography angiography represent novel and non-invasive diagnostic techniques that allow a detailed and quantitative analysis of retinal and vascular features.

The study evaluates the changes in optical coherence tomography and optical coherence tomography angiography parameters at baseline and after three monthly injections of Bevacizumab in exudative AMD.

ELIGIBILITY:
Inclusion Criteria:

* age older than 50 years, diagnosis of exudative age-related macular degeneration, treatment-naïve with Bevacizumab for exudative age-related macular degeneration.

Exclusion Criteria:

* age younger than 50 years, diagnosis of exudative macular degeneration due to other causes, previous treatments before Bevacizumab for exudative age-related macular degeneration.

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The participans were older than 50 years with diagnosis of exudative age-relative macular degeneration. They did not present other ophthalmological disease and did not receive previous treatment before Bevacizumab.
Sampling Method: Non-Probability Sample
Enrollment: 38 (Actual)
Dates: Start 2017-01-25 (Actual); Primary Completion 2017-10-25 (Actual); Study Completion 2017-10-30 (Actual)

PRIMARY OUTCOMES:
Study of retinal structural features in exudative age-related macular degeneration after intravitreal injections of Bevacizumab | three months
  The effectiveness of Bevacizumab injections for treating exudative age-related macular degeneration using optical coherence tomography. The parameters analyzed by optical coherence tomography: Central Macular Thickness and Subfoveal Choroidal thickness (microns).
Study of retinal vascular features in exudative age-related macular degeneration after intravitreal injections of Bevacizumab | three months
  The effectiveness of Bevacizumab injections for treating exudative age-related macular degeneration using optical coherence tomography angiography. The parameters analyzed by optical coherence tomography angiography were: retinal and choriocapillaris vessel density (%).

CONTACTS AND LOCATIONS:
Overall Officials: Gilda Cennamo, MD, Principal Investigator — Federico II University
Locations (1):
- University of Naples "Federico II", Naples, Italy